CLINICAL TRIAL: NCT07278362
Title: Safety of Intramuscular Testosterone Replacement Therapy in Hypogonadal Patients With Prostate Cancer Under Active Surveillance
Brief Title: Testosterone Replacement Therapy in Hypogonadal Patients With Prostate Cancer Under Active Surveillance
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Thomas Masterson, Assistant Professor of Clinical Urology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250346
Record Dates: First submitted 2025-12-04; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Hypogonadism, Male
MeSH Terms: conditions — Prostatic Neoplasms; Eunuchism | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Testosterone cypionate (Experimental): Participants will self-inject 100mg of testosterone cypionate once per week for 12 months
  Interventions: Drug: Testosterone cypionate

INTERVENTIONS:
Drug: Testosterone cypionate — Participants will self-inject 100mg of testosterone cypionate once per week for 12 months

SUMMARY:
The purpose of this study is evaluate the safety of testosterone replacement therapy in men with newly diagnosed low-risk prostate cancer and hypogonadism on active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥ 18 years old
* Newly diagnosed with low-risk prostate cancer initially confirmed by fusion guided prostate biopsy (transrectal or trans perineal) by multiparametric MRI, and had a second confirmatory biopsy within the last 12 months
* Males diagnosed with low-risk prostate cancer undergoing active surveillance
* Two confirmatory testosterone levels <300 ng/dL (taken before 10am), with at least 24 hours and no more than 90 days between the two tests
* Symptoms of low testosterone (Aging Male's Symptoms Score >27)
* Able to obtain Testosterone medication through insurance or out-of-pocket
* Willing and able to provide written informed consent and able to comply with study requirements

Exclusion Criteria:

* Males <18 years old
* History of Testosterone Replacement Therapy (TRT) within the past year.
* Current use of TRT
* Diagnosis of Gleason score 7 (Grade Group 2) prostate cancer or higher on diagnostic or confirmatory biopsy
* PSA >10 ng/mL at baseline
* Hematocrit > 51% at baseline
* T3 or T4 disease
* Uncontrolled cardiovascular disease and sleep apnea
* History of breast cancer
* Any other condition or situation which, in the opinion of the investigator, could impact patient safety, prevent successful data collection, or reduce the likelihood of successful study participation
* Unable or unwilling to obtain Testosterone medication through insurance or out-of-pocket
* Unable or unwilling to provide informed consent or comply with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Disease Progression Within 12 Months After Initiating TRT | 12 months
  Disease progression is defined as either (1) an increase in prostate cancer grade group on biopsy or (2) conversion from active surveillance to active treatment (e.g., surgery, radiation, or systemic therapy). The proportion of participants who meet either criterion within 12 months of initiating testosterone replacement therapy (TRT) will be reported.

SECONDARY OUTCOMES:
Mean Change in Serum PSA Levels (ng/mL) from Baseline to 12 Months | Baseline, 12 Months
  The mean change in serum PSA levels (ng/mL) will be measured at baseline and 12 months after initiation of TRT. PSA levels will be assessed using a standardized immunoassay. The mean change in PSA level will be used to evaluate clinical outcomes related to TRT.
Change in Total Testosterone Levels (ng/dL) from Baseline to 12 Months | Baseline, 12 Months
  The mean change in serum total testosterone (ng/dL) will be measured at baseline and 12 months after initiation of TRT. Total testosterone levels will be assessed using a standardized immunoassay. The mean change in total testosterone level will be used to evaluate clinical outcomes related to TRT.
Mean Change in Hematocrit Levels (%) from Baseline to 12 Months | Baseline, 12 Months
  The mean change in hematocrit levels (%) will be measured from baseline and 12 months after initiation of TRT. Hematocrit levels will be assessed using a standardized immunoassay. The mean change in hematocrit level will be used to evaluate clinical outcomes related to TRT.
Mean Change in Prostate Volume (mL) as measured by mpMRI from Baseline to 12 Months | Baseline, 12 Months
  The mean change in prostate volume (mL) will be measured at baseline and 12 months after initiation of TRT. Prostate volume will be calculated from T2-weighted mpMRI images using standardized volumetric analysis techniques. The mean change in volume will be used to evaluate clinical outcomes related to TRT.
Mean Change in EPIC-26 Scores from Baseline to 12 Months | Baseline, 12 Months
  Quality of life will be assessed using the EPIC-26 questionnaire at baseline and 12 months. Scores range from 0 to 100, with higher scores indicating better health-related quality of life. The mean change in scores will be used to evaluate patient-reported outcomes related to TRT.
Mean Change in SF-12 Scores from Baseline to 12 Months | Baseline, 12 Months
  Quality of life will be assessed using the SF-12 questionnaire at baseline and 12 months. The measure includes items assessing physical and mental functioning and yields two scores for these two components of quality of life. These final scores are norm-based, meaning a score of 50 represents the US population average, with a standard deviation of 10. Scores higher than 50 indicate better health status, while scores lower than 50 suggest worse health status The mean change in scores will be used to evaluate patient-reported outcomes related to TRT.
Mean Change in Aging Male's Symptoms Score (AMS) from Baseline to 12 Months | Baseline, 12 Months
  Quality of life will be assessed using the Aging Male's Symptoms Score (AMS) at baseline and 12 months. Scores range from 17 to 85, with higher scores indicating more severe symptoms. The mean change in scores will be used to evaluate symptom improvement associated with TRT.
Progression-Free Survival (PFS) from Baseline to 5 Years | Baseline to 5 Years
  Elapsed time from treatment initiation until disease progression, conversion to active treatment, or death from any cause. Median PFS, if attained, will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Masterson, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Desai Sethi Urology Institute, Miami, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida

IPD SHARING:
Plan to Share IPD: No